CLINICAL TRIAL: NCT00003773
Title: Phase I Study of Escalating Doses of IM-862 in Patients With Ovarian Cancer
Brief Title: IM-862 in Treating Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066900 (5O-98-4); LAC-USC-5O984; NCI-G99-1503
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oglufanide disodium

SUMMARY:
RATIONALE: IM-862 may stop the growth of ovarian cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of IM-862 in treating patients who have recurrent ovarian cancer after treatment with chemotherapy and surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of IM-862 administered intranasally in patients with recurrent ovarian cancer. II. Determine the toxicity of this regimen in this patient population. III. Obtain preliminary data regarding the efficacy of this drug in these patients. IV. Evaluate the effect of this drug in serum levels of vascular endothelial growth factor and transforming growth factor in this population.

OUTLINE: This is a dose escalation study. Patients receive IM-862 intranasally daily. Treatment continues for 6 months in the absence of unacceptable toxicity or disease progression. At the physician's discretion, further treatment may be given if the patient is still responding after 6 months of treatment. The dose of IM-862 is escalated in cohorts of 10-20 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 10 or 5 of 20 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 20-70 evaluable patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent ovarian cancer Failed or relapsed after cytoreductive surgery followed by a platinum-based chemotherapy regimen Measurable or evaluable disease Recurrent disease manifested by isolated increased levels of CA-125 and no other evaluable disease eligible if CA-125 is at least 100

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) ALT and/or AST no greater than 2.5 times ULN Renal: Creatinine no greater than 2 times ULN Neurological: No evidence of moderate peripheral neuropathy greater than grade 1 Other: Not pregnant Fertile patients must use effective contraception No medical, social, or psychological factors interfering with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior IM-862 No concurrent biologic therapy (e.g., interleukin-2 and interferons) Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy No concurrent antineoplastic cytotoxic agents Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy Surgery: See Disease Characteristics Recovered from prior surgery Other: No other concurrent investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1999-02; Primary Completion 2000-07 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States